CLINICAL TRIAL: NCT02748174
Title: Protective Headache Factors for Migraineurs and Postconcussive Headache Patients: Are Behavioral Strategies Effective? A Naturalistic Study
Brief Title: Protective HA Factors
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: screening survey data was not correctly collected; Study halted prematurely
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-01055
Record Dates: First submitted 2016-04-19; First posted 2016-04-22 (Estimated); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Post Concussive Headache
Keywords: Migraine; Curelator
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Episodic Migraine group (Experimental): 100 patients with chronic or episodic migraine
  Interventions: Behavioral: Audio Files
- Chronic Migraine Group (Experimental): 100 patients with chronic or episodic migraine
  Interventions: Behavioral: Audio Files
- Post concussive Headache Group (Experimental): 75 patients
  Interventions: Behavioral: Audio Files

INTERVENTIONS:
Behavioral: Audio Files — Patients will be given a link to download audio files. They consist of breathing techniques, imaging, progressive relaxation, and more. Patients will be asked to perform 20 minutes of relaxation therapy at least 3 times per week. Patients will record their headache frequency and intensivy, in addition to other symptoms, and the frequency of practiving the behavioral therapy using Curelator Headache.

SUMMARY:
This is a naturalistic study of 100 migraineurs and 75 post concussive headache patients who will be asked to record their headaches, medications, sleep and other behaviors in a smartphone app called Curelator. The software was developed to identify possible headache triggers. We seek to determine whether there might be protective headache factors. Patients will be given audio files with relaxation therapies. We seek to understand whether this self relaxation therapy and/or traditional evidence based behavioral treatment recommended during a patient visit is protective against migraine attacks.

DETAILED DESCRIPTION:
Patients will be given a link to audio files on dropbox which they can download onto their smartphone. They consist of breathing techniques, imaging, progressive relaxation, and more. Patients will be asked to perform 20 minutes of relaxation therapy at least 3 times a week. Patients will record their headache frequency and intensity, in addition to other symptoms, and the frequency of practicing the behavioral therapy using Curelator Headache. ™ Curelator Inc. (Cambridge USA) has developed a proprietary, non-pharmaceutical, digital platform, called Curelator Headache,™ to collect daily data, identify trigger-attack associations and propose 'tests' of trigger modification.

The Curelator approach requires high quality data from the individual, entered on a daily basis. Compliance is expected to be enhanced because the study if being offered by the individual's healthcare provider.

This a pilot study of an initial 90 days use of a digital platform to identify potential migraine protective factors (Curelator Headache™) in subjects with physician-diagnosed episodic or chronic migraine or post-concussive headache. Subjects are recruited to Curelator Headache use by a physician and enter data each day. The baseline period (90 days) is followed by a test period (90 days) during which, under Curelator guidance, subjects make one or more modifications to their behaviors based on the data from the 90 day period.

The study will include up to 100 patients with chronic or episodic migraine and 75 patients with postconcussive headache. At clinics, investigators will offer participation to consecutive migraine patients with 6-20 headache days a month and to consecutive concussion patients complaining of headache more than 1 month post concussive event.

ELIGIBILITY:
Inclusion Criteria:

* Male or female reporting at least 6 month history of episodic or chronic migraine with 6-20 headache days a month
* Age: 18-65 years
* Age of onset of migraine was <age 50
* Able to give informed consent/assent
* Sufficiently fluent in English to be able to use the English language version of Curelator Headache (no translations available).
* Has ownership of or reliable access to iPhone or (mini) iPad running iOS 7 or higher
* Able to give written informed consent (adults), or, for adolescents, has a parent/caregiver who can give informed consent and adolescent is able to give assent.
* Willing to use Curelator Headache for at least 3 months and to comply with study procedures.
* In the Investigator's opinion, there is no reason to believe that Curelator Headache use would pose any risk to the patient.

Exclusion Criteria:

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Number of completers (assessment of adherence) | 90 Days
Number of days with migraine and other headache | 90 Days
Number of migraine headaches | 90 Days
Number of significant trigger/warning sign - migraine attack associations | 90 Days
  This will be analyzed by means of univariate Cox Proportional Hazards (PH) models. At the end of the study period (Day 90) significant trigger factors (HR/RR>1 and p-value ≤ 0.05) will be identified for each individual: the number and percentage of subjects with at least one significant relationship between a trigger and occurrence of migraine attacks and the number of trigger-migraine attack significant relationships per individual will be estimated by means of descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Mia Minen, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University Langone Medical Center, New York, New York, United States